CLINICAL TRIAL: NCT01044173
Title: Assessment of Patients With Nontraumatic Acute Abdominal Pain With Plain MR of the Abdomen - a Comparison With CT
Brief Title: Plain Magnetic Resonance (MR) in the Assessment of Patients With Acute Abdomen
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Jens Maier, overlæge, radiologisk afdeling, Køge sygehus, Zealand University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N-20090033
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Acute Abdomen
Keywords: acute abdomen; CT; MRI; fast imaging
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MR scan — axial and coronal free breathing HASTE sequences 3D T1 weighted gradient echo breathhold

SUMMARY:
At present, CT is the gold standard in the assessment of patients with acute abdomen. Yet, one CT of the abdomen exposes patients to a radiation dose equivalent to several years of background radiation. MR can be expected to yield the same information without ionizing radiation, but tends to be more time consuming. In this study, patients with nontraumatic acute abdominal pain referred to CT of the abdomen by the department of surgery will also have performed an additional MR scan covering the entire abdomen with few fast imaging sequences in approximately 15min. CT is the diagnostic test. The MR scan is only used for scientific purposes. It will be evaluated by a radiologist blinded for the results of the CT scan. Fourteen days after admission, a final diagnosis is established based on clinical, peroperative, pathological and lab. findings. The performance of CT and MR will then be compared. The investigators hypothesize that MR can provide a diagnostic accuracy comparable to CT.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age > 18 years old
* Nontraumatic acute abdomen
* Weight < 120kg
* Can keep apnoea for 15s
* Surgeon in charge considers patient fit for participation in study

Exclusion Criteria:

* Contraindications of MRI
* Suspicion of acute vascular disease
* Severe cardial or pulmonal insufficiency
* Pregnancy
* Untreated psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy of CT vs. MR | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jørgensen, MD, Principal Investigator — Zealand University Hospital; Jens Maier, MD, Study Director — Zealand University Hospital
Locations (1):
- Koege Sygehus, Koege, Denmark

REFERENCES:
- [Background] Stoker J. Magnetic resonance imaging and the acute abdomen. Br J Surg. 2008 Oct;95(10):1193-4. doi: 10.1002/bjs.6378. No abstract available. PMID 18763236